CLINICAL TRIAL: NCT00003152
Title: Marrow-Ablative Chemo-Radiotherapy and Autologous Stem Cell Transplantation Followed by Interferon-Alpha Maintenance Treatment Versus Interferon-Alpha Maintenance Treatment Alone After a Chemotherapy-Induced Remission in Patients With Stages III or IV Follicular Non-Hodgkin's Lymphoma. A Prospective, Randomized, Phase III Clinical Trial.
Brief Title: Chemotherapy Plus Interferon Alfa Alone or With Radiation Therapy and Peripheral Stem Cell Transplantation in Treating Patients With Stage III or Stage IV Follicular Non-Hodgkin's Lymphoma
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: low accrual
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Collaborators: Lymphoma Trials Office (Other); Stichting Hemato-Oncologie voor Volwassenen Nederland (Other)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: EORTC-20963; EORTC-20963; BNLI-EORTC-20963; HOVON-35
Record Dates: First submitted 1999-11-01; First posted 2004-08-02 (Estimated); Last update posted 2012-07-02 (Estimated); Status verified 2012-06

CONDITIONS: Lymphoma
Keywords: stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Follicular | interventions — Filgrastim; Interferon-alpha; Cyclophosphamide; Prednisone; Vincristine; Peripheral Blood Stem Cell Transplantation; Radiotherapy

INTERVENTIONS:
Biological: filgrastim
Biological: recombinant interferon alfa
Drug: cyclophosphamide
Drug: prednisone
Drug: vincristine sulfate
Procedure: autologous bone marrow transplantation
Procedure: bone marrow ablation with stem cell support
Procedure: peripheral blood stem cell transplantation
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Interferon alfa may interfere with the growth of cancer cells. Radiation therapy uses high-energy x-rays to damage cancer cells. Peripheral stem cell transplantation may allow the doctor to give higher doses of chemotherapy drugs and radiation therapy and kill more cancer cells.

PURPOSE: Randomized phase III trial to compare the effectiveness of combination chemotherapy followed by interferon alfa alone or combination chemotherapy plus radiation therapy and peripheral stem cell transplantation in treating patients who have previously untreated stage III or stage IV follicular non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES: I. Compare the progression free and overall survival, toxicity, and mortality of marrow ablative chemo/radiotherapy in addition to peripheral blood stem cell transplantation and interferon alfa maintenance therapy versus interferon alfa maintenance therapy alone in patients with follicular non-Hodgkin's lymphoma.

OUTLINE: This is a randomized study. All patients receive 8 courses of cyclophosphamide/vincristine/prednisone (CVP) chemotherapy. Cyclophosphamide and vincristine IV are given on day 1, along with oral prednisone on days 1-5. Courses are repeated every 3 weeks. Patients are randomized to receive one of two treatments 4 weeks after completion of CVP chemotherapy if a partial or complete response is achieved and there are less than 15% monoclonal B-lymphocytes in the bone marrow. Patients randomized to arm I receive interferon alfa subcutaneously 3 times per week for a maximum of 3 years. Patients randomized to arm II receive cyclophosphamide IV followed by subcutaneous filgrastim (granulocyte colony-stimulating factor; G-CSF). Leukapheresis begins after leukocyte, platelet, and CD34+ levels recover and lasts 3-4 hours on 2-3 consecutive days. If an insufficient number of stem cells are collected from the peripheral blood, bone marrow harvesting is performed. After stem cell collection, a conditioning regimen consisting of cyclophosphamide IV on days -4 and -3 and total body irradiation on day -1 is administered. Stem cells are infused on day 0. If granulocyte and platelet counts recover within 8 weeks, patients receive interferon alfa maintenance therapy as in arm I. Patients are followed every 4 months until death.

PROJECTED ACCRUAL: A total of 469 patients will be accrued for this study within 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Previously untreated follicular stage III or IV non-Hodgkin's lymphoma At least one measurable mass

PATIENT CHARACTERISTICS: Age: 18 to 65 Performance status: WHO 0-2 Life expectancy: Not specified Hematopoietic: Not specified Hepatic: Alkaline phosphatase and bilirubin less than 2.5 times upper limit of normal (ULN) (unless clearly related to NHL) Renal: Creatinine and BUN less than 2.5 times ULN (unless clearly related to NHL) Cardiovascular: No severe cardiac disease (e.g. severe heart failure requiring treatment or cardiac ejection fraction less than 45%) Neurologic: No neurologic disease Pulmonary: No pulmonary disease Other: Not pregnant No prior malignancies except nonmelanoma skin cancer or carcinoma in situ of the cervix Not HIV positive No psychiatric or metabolic disease

PRIOR CONCURRENT THERAPY: See Disease Characteristics No concurrent immunotherapeutic drugs, chemotherapy, or radiotherapy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 469 (Estimated)
Dates: Start 1997-03; Primary Completion 1999-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anton Hagenbeek, MD, PhD, Study Chair — UMC Utrecht; Robert Marcus, MD, Study Chair — Cambridge University Hospitals NHS Foundation Trust
Locations (2):
- Academisch Ziekenhuis Utrecht, Utrecht, Netherlands
- Addenbrooke's NHS Trust, Cambridge, England, United Kingdom